CLINICAL TRIAL: NCT01048099
Title: Use of the PRO Onc Assay to Assess HER2 Overexpression and Activation in Patients With Metastatic Breast Cancer Whose Tumors Are HER2-Negative by Standard FISH Testing
Brief Title: Use of PRO Onc Assay to Assess HER2 in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Prometheus Laboratories (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 166
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastatic; PRO Onc Assay; FISH Testing; HER Negative; HER Overexpression; HER Activation
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Therapeutics; Blood Specimen Collection; Biopsy, Fine-Needle; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRO Onc Assay and Treatment (Experimental): Blood specimens tested for circulating tumor cells followed by systemic treatment based on assay results with either trastuzumab or pertuzumab
  Interventions: Procedure: PRO Onc Assay and Treatment; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Procedure: PRO Onc Assay and Treatment — Patients with HER2-negative metastatic breast cancer will be identified, and blood specimens will be obtained from each participant. The PRO Onc Assay will be performed on CTCs isolated from these specimens. When clinically indicated, fine needle aspiration biopsy will also be obtained and submitted for the PRO Onc Assay.
  Other Names: blood draw; fine needle aspiration; circulating tumor cells
Drug: Trastuzumab — 8 mg/kg IV loading dose, followed by 6 mg /kg IV every 3 weeks until progressive disease or unacceptable toxicity with evaluations performed every 8 weeks
  Other Names: Herceptin
Drug: Pertuzumab — 840 mg IV loading dose, followed by 420 IV every 3 weeks until progressive disease or unacceptable toxicity with evaluations performed every 8 weeks
  Other Names: Perjeta

SUMMARY:
This trial will evaluate the clinical significance of the PRO Onc assay and will assess the efficacy of HER2-targeted therapy in patients with HER2-negative breast cancer who have been identified as having HER2 overexpression/activation by the PRO Onc Assay.

DETAILED DESCRIPTION:
This two-part trial is designed to evaluate the clinical significance of the PRO Onc assay when used in patients with metastatic HER2-negative breast cancer. The first part of this study will determine the incidence of HER overexpression/activation, as determined by the PRO Onc assay, in patients previously judged to have HER2-negative breast cancer by FISH analysis. Blood specimens will be obtained from patients with HER2-negative breast cancer; CTCs will then be isolated and tested for HER2 overexpression/activation using the PRO Onc Assay. When clinically indicated, fine needle aspiration biopsy will also be obtained and submitted for the PRO Onc Assay. If the incidence of HER2 overexpression/activation, as determined by the PRO Onc Assay, is >10%, the study will proceed to Part 2. Part 2 of this study will assess the efficacy of HER2-targeted therapy in a group of patients with HER2-negative breast cancer who are identified as having HER2 overexpression/activation by the PRO Onc Assay. Patients will be treated with either trastuzumab or pertuzumab. Patients who progress during the first 8 weeks will have HER2-targeted treatment discontinued and will be removed from study. After 8 weeks, patients who have stable disease will be allowed to add chemotherapy to HER2-targeted therapy. Patients who have an objective response to single-agent, HER2-targeted therapy after 8 weeks will continue single-agent therapy.

ELIGIBILITY:
Inclusion Criteria:

Part I

1. Women with HER2-negative breast cancer, as defined by FISH testing. (FISH testing may have been performed on the primary tumor, or subsequently on a biopsy of a metastatic lesion.)
2. Patients should be currently receiving chemotherapy, or scheduled to start chemotherapy (second-line or subsequent), for HER2-negative metastatic breast cancer.
3. To begin protocol treatment, patients must have progressed after at least 1 previous chemotherapy regimen for metastatic breast cancer.
4. Patients who are ER/PR positive or negative are eligible. ER/PR positive patients should be refractory to hormonal therapy, or not good candidates for hormonal therapy due to clinical features.
5. ECOG performance status of 0, 1 or 2.
6. Adequate recovery from recent surgery; ≥ 1 week must have elapsed from the time of a minor surgery; ≥ 4 weeks must have elapsed from the time of a major surgery.
7. Patients must have measurable disease per RECIST criteria.
8. Laboratory values as follows: Absolute neutrophil count (ANC) ≥1500/μL Hemoglobin (Hgb) ≥10 g/dL Platelets ≥100,000/L AST or ALT and alkaline phosphatase (ALP) must be <2.5 x ULN, or <5 x ULN in patients with liver metastases. Total bilirubin <1.5 x the institutional ULN Serum creatinine <1.5 x institutional ULN or calculated creatinine clearance ≥45 mL/min

   Patients from Part 1 who have HER2 overexpression/activation identified by the PRO Onc Assay may enter the treatment portion of Part 2, if they meet all Part 2 eligibility criteria.
9. Life expectancy of ≥ 12 weeks.
10. Patient must be accessible for treatment and follow-up.
11. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.

Part II

1. Women with HER2-negative breast cancer, as defined by FISH testing. (FISH testing may have been performed on the primary tumor, or subsequently on a biopsy of a metastatic lesion.)
2. Patients should be currently receiving chemotherapy, or scheduled to start chemotherapy, for HER2-negative metastatic breast cancer.
3. Patients who are ER/PR positive or negative are eligible. ER/PR positive patients should be refractory to hormonal therapy, or not good candidates for hormonal therapy due to clinical features.
4. ECOG performance status of 0, 1 or 2.
5. Adequate recovery from recent surgery; ≥ 1 week must have elapsed from the time of a minor surgery; ≥ 4 weeks must have elapsed from the time of a major surgery.
6. Patients must have measurable disease per RECIST criteria.
7. Laboratory values as follows:

   * Absolute neutrophil count (ANC) ≥1500/μL
   * Hemoglobin (Hgb) ≥10 g/dL
   * Platelets ≥100,000/uL
   * AST or ALT and alkaline phosphatase (ALP) must be <2.5 x ULN, or <5 x ULN in patients with liver metastases.
   * Total bilirubin <1.5 x the institutional ULN
   * Serum creatinine <1.5 x institutional ULN or calculated creatinine clearance ≥45 mL/min
8. Life expectancy of ≥ 12 weeks.
9. Patient must be accessible for treatment and follow-up.
10. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.
11. Patients who are eligible for HER2-targeted treatment will begin this treatment at the first time a treatment change is necessary (i.e. at the next progression of metastatic breast cancer). This may occur immediately after PRO Onc assay results are received, or may be several months later, for patients responding well to their current chemotherapy.
12. Patients must continue to meet all inclusion and exclusion criteria for the Part 2 screening population at the time they are ready to start HER2-targeted treatment.
13. Ejection fraction ≥ 50%, as measured by echocardiogram (ECHO) or MUGA.

Exclusion Criteria:

Part I:

1. Patients currently responding to hormonal therapy.
2. Previous treatment with any HER2-targeted agent.
3. Patients with meningeal metastases.
4. Patients who are not considered likely candidates for subsequent therapy after next progression of metastatic breast cancer.
5. Women who are pregnant or lactating.
6. Patients with New York Heart Association class II or greater congestive heart failure.
7. Any of the following ≤6 months prior to starting study treatment:

   * myocardial infarction;
   * severe unstable angina;
   * ongoing cardiac dysrhythmia
8. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements.
9. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
10. Use of any non-approved or investigational agent ≤ 30 days of administration of the first dose of study drug. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.

Part II

1. Patients currently responding to hormonal therapy.
2. Previous treatment with any HER2-targeted agent.
3. Patients with meningeal metastases.
4. Patients with active brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if there is no evidence of central nervous system (CNS) disease progression, and at least 4 weeks have elapsed since treatment. Ideally, patients should not still require use of seizure medication or steroids.
5. Patients who are not considered likely candidates for subsequent therapy after next progression of metastatic breast cancer.
6. Women who are pregnant or lactating.
7. Patients with New York Heart Association class II or greater congestive heart failure.
8. Any of the following ≤6 months prior to starting study treatment:

   * myocardial infarction;
   * severe unstable angina;
   * ongoing cardiac dysrhythmia.
9. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements.
10. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
11. Use of any non-approved or investigational agent ≤ 30 days of administration of the first dose of study drug. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
12. Past or current history of neoplasm other than the entry diagnosis with the exception of treated non-melanoma skin cancer or carcinoma in situ of the cervix, or other cancers cured by local therapy alone and a DFS ≥5 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (7):
- United States (7):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Virginia Cancer Institute, Richmond, Virginia

REFERENCES:
- [Derived] Hainsworth JD, Murphy PB, Alemar JR, Daniel BR, Young RR, Yardley DA. Use of a multiplexed immunoassay (PRO Onc assay) to detect HER2 abnormalities in circulating tumor cells of women with HER2-negative metastatic breast cancer: lack of response to HER2-targeted therapy. Breast Cancer Res Treat. 2016 Nov;160(1):41-49. doi: 10.1007/s10549-016-3969-7. Epub 2016 Sep 8. PMID 27632289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pts with HER2-negative, metastatic breast cancer were enrolled. Blood was collected to perform the PRO Onc Circulating Tumor Cell (CTC). Pts without CTCs present were taken off-study. Following the assay, pts without detected HER2 overexpression/activation were taken off-study. Of the remaining pts, those FISH-positive for HER2 came off-study.
Period: Patients Enrolled and Blood Collected
Arm/Group | All Patients
Started | 283 (Patients enrolled)
Completed | 226 (Patients with circulating tumor cells (CTCs))
Not Completed | 57
Not completed — Patients without circulating tumor cells | 57
Period: Patients Evaluated by PRO Onc Assay
Arm/Group | All Patients
Started | 226 (Patients with CTCs who were evaluated by PRO Onc Assay)
Completed | 24 (Patients evaluated by PRO Onc Assay with HER2 overexpression/activation detected)
Not Completed | 202
Not completed — Patients with no HER2 abnormality | 202
Period: Pts w/ HER2 Overexpression/Activation
Arm/Group | All Patients
Started | 24 (Patients with detected HER2 activation and/or overexpression)
Completed | 14 (Patients who proceeded to treatment)
Not Completed | 10
Period: Treatment Per Protocol
Arm/Group | All Patients
Started | 14
Completed | 0 (Patients continued treatment until disease progression or coming off-study for any other reason)
Not Completed | 14

BASELINE CHARACTERISTICS:
Population: Excludes patients with no circulating tumor cells for the PRO Onc Assay
Groups:
- Patients Treated: Patients who received study treatment
Arm/Group | Patients Treated
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 65 [47 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Secondary Outcome: Part 1: The Incidence of HER2 Overexpression/Activation as Measured by the PRO Onc Assay
Description: Includes patients with HER2-negative metastatic breast cancer (MBC) as determined by FISH testing.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | All Patients Evaluated by PRO Onc Assay
Number analyzed (Participants) | 226
participants
  HER2 overexpressed | 11
  HER2 activated | 10
  HER2 overexpressed and activated | 3
  No HER2 overexpression/activation detected | 202

2. Primary Outcome: Part II: Objective Response Rate of HER2-negative Metastatic Breast Cancer (by FISH Testing)
Description: The percentage of HER2-negative metastatic breast cancer (MBC) patients having an objective benefit from treatment per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Includes patients with HER2 overexpression/activation as detected by PRO Onc Assay.
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Patients Treated
Number analyzed (Participants) | 14
percentage of participants | 7

3. Secondary Outcome: Part I: The Incidence of Isolation of Circulating Tumor Cells (CTCs) From Blood Specimens
Description: Percentage of HER2-negative MBC patients (identified by FISH testing) having CTCs present in blood specimens.
Time Frame: 12 months
Population: Includes all patients with blood drawn and analyzed for CTCs
Measure: Number; unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 283
percentage of participants | 80

4. Primary Outcome: Part II: Objective Response Rate of Trastuzumab Therapy
Description: The percentage of patients having an objective benefit from treatment per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Includes patients with HER2 overexpression as identified by the PRO Onc Assay.
Time Frame: 18 months
Population: Includes patients with HER2 overexpression detected by the PRO Onc Assay
Measure: Number; unit: percentage of participants
Arm/Group | Patients Treated
Number analyzed (Participants) | 10
percentage of participants | 10

5. Primary Outcome: Part II: Objective Response Rate of Pertuzumab Therapy
Description: The percentage of patients with HER2 activation (no overexpression) as identified by the PRO Onc Assay who experience an objective benefit from treatment, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Population: Includes patients with only HER2 activation (no overexpression) as detected by the PRO Onc Assay
Measure: Number; unit: percentage of participants
Arm/Group | Patients Treated
Number analyzed (Participants) | 4
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: 18 Months
Groups:
- All Treated Patients: Includes all patients with HER2 overexpression/activation (as identified by the PRO Onc Assay) who received study treatment
Arm/Group | All Treated Patients
Serious Adverse Events (participants affected / at risk) | 5/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Patients (N=14)
General disorders and administration site conditions - Other, disease progression (General disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Infections and infestations - Other, pneumonia (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Patients (N=14)
Fatigue (General disorders) | 7
Infusion related reaction (General disorders) | 4
Urinary Tract Infection (Infections and infestations) | 4
Anorexia (Metabolism and nutrition disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Allergic reaction (Immune system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Edema (General disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anxiety (Psychiatric disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Fever (General disorders) | 1
Headache (Nervous system disorders) | 1
Renal and urinary disorders - Other, hydronephrosis (Renal and urinary disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hepatobiliary disorders - Other, liver dysfunction (Hepatobiliary disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Skin infection (Infections and infestations) | 1
Dysgeusia (Nervous system disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, thoracic pain (Respiratory, thoracic and mediastinal disorders) | 1
Platelet count decreased (Investigations) | 1
Urinary frequency (Renal and urinary disorders) | 1
Weight loss (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites